CLINICAL TRIAL: NCT00263172
Title: Weight Loss on the Web: A Pilot Study Comparing a Commercial Website to a Structured Behavioral Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS# 03-022
Record Dates: First submitted 2005-12-05; First posted 2005-12-07 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2005-12

CONDITIONS: Obesity; Diet Therapy; Weight Loss
Keywords: internet; weight management; behavior therapy; self-help; commercial program; obesity
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: behavior modification for weight loss

SUMMARY:
The primary purpose of this study was to compare weight loss achieved through a behavioral online intervention vs. a commercial self-help website. The investigators hypothesized that there would be no difference in weight loss between groups.

DETAILED DESCRIPTION:
Obesity has reached epidemic proportions in the United States. Novel approaches are needed to address this issue on a broad scale. The internet holds promise as a way to disseminate effective weight loss strategies. The primary purpose of this study was to compare weight loss achieved through a behavioral online intervention vs. a commercial self-help website. A second aim was to evaluate the utilization of web components and their relationship to weight loss between groups and within groups in order to determine what aspects of web usage correlate to weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 39.9 kg/m2
* 18 or older

Exclusion Criteria:

* Planned to move within 1 year
* Planned a pregnancy within 1 year
* Take medications with weight implications
* Unable to exercise moderately
* Participating in another weight loss program
* Lacked minimum computer requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Study Completion 2005-03

PRIMARY OUTCOMES:
weight change

SECONDARY OUTCOMES:
social influence components
eating behavior
web usage correlation to weight change

CONTACTS AND LOCATIONS:
Overall Officials: Doris E Ogden, MS, LCMHC, Study Director — University of Vermont
Locations (1):
- Behavioral Weight Management Program/Univ of Vermont, Burlington, Vermont, United States